CLINICAL TRIAL: NCT01508819
Title: Impact on Mid-term Mortality of Guidelines for ICU Admission of Elderly Patients Arriving in Emergency Departments: a Cluster Randomized Controlled Trial
Brief Title: Impact on Mid-term Mortality of Guidelines for ICU Admission of Elderly Patients Arriving in Emergency Departments
Acronym: ICECUBII
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K100103
Record Dates: First submitted 2011-12-09; First posted 2012-01-12 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Elderly Patients Visiting the Emergency Department
Keywords: Patients over 75; acute pathology; ICU admission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Guidelines for ICU admission of elderly patients arriving in Emergency Departments with a life threatening conditions
  Interventions: Other: recommendations to admit to ICU all the patients included
- 2: no intervention

INTERVENTIONS:
Other: recommendations to admit to ICU all the patients included — recommendations to emergency and ICU physicians to admit to ICU all the patients included in the trial
  Groups: 1

SUMMARY:
Admitting a very elderly patient to the Intensive Care Unit (ICU) is one of the most difficult clinical challenges in medicine. There are few data to help guide clinicians in this area: estimates of the benefits of ICU admission, especially in the very elderly, are sparse. Rates of ICU admission of very elderly thus vary widely by hospitals.

The ICE-CUB1 (PHRC AOR 03 035) project has studied the ICU admission decision process of patients over 80 arriving in Emergency Departments (ED) with conditions that potentially warrant ICU admission and their outcome six months after ED visit. Overall rate of patients deemed eligible for ICU admission was of 12% (Garrouste et al. Crit Care Med 2009) but ranged from 5% to 38% across the participating centers. This variability persisted after adjustment for patients' characteristics (MOR 2.25, 1.60-3.58; hospital-related variance 18%). The analysis also revealed that high functional status prior to ICU visit, good nutritional status as assessed by an emergency physician and the absence of cancer were of good prognosis for outcome six months after ED visit. Only 23% of patients visiting the ED with a life-threatening condition and all positive prognostic factors mentioned above were admitted to an ICU in the ICE-CUB1 study.

Hypothesis Elderly patients visiting the ED with a life-threatening condition, high functional status prior to ICU visit, good nutritional status as assessed by an emergency physician and no cancer will potentially benefit from ICU care and should thus be admitted.

Main objective Determine whether a strategy consisting of recommendations of ICU admission of all patients over 75 visiting the ED with a life threatening condition, no cancer, good functional and nutritional status prior to ED visit decreases the mortality of these patients six months after ED visit.

Secondary objective : Assess the impact of the strategy on:

* In-hospital mortality
* Rate of ICU admission
* Place of living and quality of life six months after ED visit

Primary outcome :Mortality six months after ED visit Secondary outcomes

* In-hospital mortality
* ICU admission
* Change in functional status six months after ED visit
* institutionalization
* Quality of life six months after ED visit

DETAILED DESCRIPTION:
Admitting a very elderly patient to the Intensive Care Unit (ICU) is one of the most difficult clinical challenges in medicine. There are few data to help guide clinicians in this area: estimates of the benefits of ICU admission, especially in the very elderly, are sparse. Rates of ICU admission of very elderly thus vary widely by hospitals.

The ICE-CUB1 (PHRC AOR 03 035) project has studied the ICU admission decision process of patients over 80 arriving in Emergency Departments (ED) with conditions that potentially warrant ICU admission and their outcome six months after ED visit. Overall rate of patients deemed eligible for ICU admission was of 12% (Garrouste et al. Crit Care Med 2009) but ranged from 5% to 38% across the participating centers. This variability persisted after adjustment for patients' characteristics (MOR 2.25, 1.60-3.58; hospital-related variance 18%). The analysis also revealed that high functional status prior to ICU visit, good nutritional status as assessed by an emergency physician and the absence of cancer were of good prognosis for outcome six months after ED visit. Only 23% of patients visiting the ED with a life-threatening condition and all positive prognostic factors mentioned above were admitted to an ICU in the ICE-CUB1 study.

Hypothesis Elderly patients visiting the ED with a life-threatening condition, high functional status prior to ICU visit, good nutritional status as assessed by an emergency physician and no cancer will potentially benefit from ICU care and should thus be admitted.

Main objective Determine whether a strategy consisting of recommendations of ICU admission of all patients over 75 visiting the ED with a life threatening condition, no cancer, good functional and nutritional status prior to ED visit decreases the mortality of these patients six months after ED visit.

Secondary objective : Assess the impact of the strategy on:

* In-hospital mortality
* Rate of ICU admission
* Place of living and quality of life six months after ED visit

Primary outcome :Mortality six months after ED visit Secondary outcomes

* In-hospital mortality
* ICU admission
* Change in functional status six months after ED visit
* institutionalization
* Quality of life six months after ED visit

Type of study Cluster stratified randomized controlled trial. Stratification criteria are existence of an acute geriatric ward, capacity of the emergency department and location of the hospital (in or out Paris area)

ELIGIBILITY:
Inclusion Criteria:

* Age over 75 years old
* At least one organ failure
* No cachexia
* No active known cancer
* Good functional status (as assessed by an ADL score > 4) or not evaluable
* Affiliated to social security

Exclusion Criteria:

* refusal

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 75 visiting the emergency department with a condition potentially warranting intensive care unit admission
Sampling Method: Probability Sample
Enrollment: 3036 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mortality six months after emergency department visit | 6 months after emergency department visit

SECONDARY OUTCOMES:
hospital mortality | up to 6 months
ICU admission rate | length of hospital stay
change in functional status | 6 months after emergency department visit
institutionalization | 6 months after emergency department visit
quality of life | 6 months after emergency department visit

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Guidet, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- ICU - Saint-Antoine Hospital, Paris, France

REFERENCES:
- [Derived] Guidet B, Leblanc G, Simon T, Woimant M, Quenot JP, Ganansia O, Maignan M, Yordanov Y, Delerme S, Doumenc B, Fartoukh M, Charestan P, Trognon P, Galichon B, Javaud N, Patzak A, Garrouste-Orgeas M, Thomas C, Azerad S, Pateron D, Boumendil A; ICE-CUB 2 Study Network. Effect of Systematic Intensive Care Unit Triage on Long-term Mortality Among Critically Ill Elderly Patients in France: A Randomized Clinical Trial. JAMA. 2017 Oct 17;318(15):1450-1459. doi: 10.1001/jama.2017.13889. PMID 28973065
- [Derived] Boumendil A, Woimant M, Quenot JP, Rooryck FX, Makhlouf F, Yordanov Y, Delerme S, Takun K, Ray P, Kouka MC, Poly C, Garrouste-Orgeas M, Thomas C, Simon T, Azerad S, Leblanc G, Pateron D, Guidet B; ICE-CUB 2 study network. Designing and conducting a cluster-randomized trial of ICU admission for the elderly patients: the ICE-CUB 2 study. Ann Intensive Care. 2016 Dec;6(1):74. doi: 10.1186/s13613-016-0161-5. Epub 2016 Jul 29. PMID 27473119